CLINICAL TRIAL: NCT04881058
Title: Post Market Clinical Follow Up Study to Collect Additional Data and Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7012-BDPM-2021
Record Dates: First submitted 2021-05-03; First posted 2021-05-11 (Actual); Results first posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Pigmentation; Wrinkle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- PicoSure Device (Experimental): The PicoSure device will be used on the face for the treatment of pigmentation and mild to moderate wrinkles.
  Interventions: Device: RF Non-Invasive Treatment

INTERVENTIONS:
Device: RF Non-Invasive Treatment — Self-controlled single-arm group using the PicoSure device.

SUMMARY:
The intended use of the PicoSure device with focus lens array used in this study is to assess images to support additional marketing claims for the treatment of pigmentation and mild to moderate wrinkles.

DETAILED DESCRIPTION:
Up to 10 subjects will be enrolled at 1 study center. Subjects will attend a screening/pretreatment visit which may be performed on the same day as the treatment visit. Subjects may receive up to 4 treatments on the face with the PicoSure device.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female 18 - 65 years of age.
* Willing to undergo treatments for pigmentation and/or mild to moderate wrinkles on the face with the PicoSure device.
* Understands and accepts obligation not to receive any other procedures on the treatment area through the length of the study.
* Understands and accepts the obligation and is logistically able to be present for all visits.
* Is willing to comply with all requirements of the study and sign the informed consent document.

Exclusion Criteria:

* Is pregnant or of childbearing potential and not using medically effective birth control, or has been pregnant in the last 3 months, currently breast feeding or planning a pregnancy during the study.
* The subject is hypersensitive to light in the near infrared wavelength region.
* The subject takes medication which is known to increase sensitivity to sunlight.
* The subject has seizure disorders triggered by light.
* The subject takes or has taken oral isotretinoin, such as Accutane®, within the last six months.
* The subject has an active localized or systemic infection, or an open wound in area being treated.
* The subject has a significant systemic illness, such as lupus, or an illness localized in area being treated.
* The subject has common acquired nevi that are predisposed to the development of malignant melanoma.
* The subject has herpes simplex in the area being treated.
* The subject is receiving or has received gold therapy.
* The subject is currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within in the area to be treated 6 months to entering this study.
* The subject has any condition or is in a situation which in the investigators opinion may put the subject at significant risk, may confound study results or may interfere significantly with the subject's participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Civiok, Study Director — Cynosure, Inc.
Locations (1):
- New Jersey Plastic Surgery, Montclair, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gupta V, Sharma VK. Skin typing: Fitzpatrick grading and others. Clin Dermatol. 2019 Sep-Oct;37(5):430-436. doi: 10.1016/j.clindermatol.2019.07.010. Epub 2019 Jul 17. PMID 31896400

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PicoSure Device
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PicoSure Device
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 5
  Hispanic | 3
  Asian | 2
FitzPatrick Skin Type [Count of Participants; unit: Participants] — Subjects were graded on a Fitzpatrick Skin Type scale from I-VI, with I representing a low melanin content, and VI representing a higher melanin content. This grading criteria/scale comes from the reference listed in the protocol section.
  Participants
    Fitzpatrick Skin Type I | 0
    Fitzpatrick Skin Type II | 4
    Fitzpatrick Skin Type III | 5
    Fitzpatrick Skin Type IV | 1
    Fitzpatrick Skin Type V | 0
    Fitzpatrick Skin Type VI | 0

OUTCOME MEASURES:

1. Primary Outcome: Correct Identification of Baseline Photographs vs. Photographs Taken 3 Months Post Last Treatment
Description: Three blinded independent reviewers will perform a photographic evaluation in which they will be asked to identify pre-treatment images when compared to post treatment images. The percentage of photographs that were correctly identified as either baseline photographs or photographs taken at the 3 month follow up will be reported. Identifying whether the photograph was taken at the baseline vs. 3 month follow up was only done at the 3 month follow up point.
Time Frame: 3 month follow up
Measure: Number; unit: % of photos correctly identified
Units Other Than Participants: photographs
Arm/Group | PicoSure Device
Number analyzed (Participants) | 10
Number analyzed (photographs) | 30
% of photos correctly identified | 80

ADVERSE EVENTS:
Time Frame: Adverse events were collected from up to 9 months from the baseline
Arm/Group | PicoSure Device
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT04881058/Prot_SAP_000.pdf